CLINICAL TRIAL: NCT02552498
Title: Post Occlusive Reactive Hyperemia on Gingiva Assessed by Laser Speckle Contrast Imaging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Semmelweis University (Other)
Responsible Party: Principal Investigator, Dr. Vag Janos, associate professor, Semmelweis University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2/2013
Record Dates: First submitted 2015-09-15; First posted 2015-09-17 (Estimated); Last update posted 2018-04-19 (Actual); Status verified 2018-04

CONDITIONS: Ischemia
MeSH Terms: conditions — Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- vertical (Experimental): Strangulation is applied on the the buccal side of the attached gingiva, parallel to the long axis of tooth 12, at the distal third of the tooth.
  Interventions: Procedure: strangulation
- horizontal (Experimental): Strangulation is applied on the buccal side of the attached gingiva, perpendicular to the long axis of the tooth 12, 2 mm far from the gingival margin.
  Interventions: Procedure: strangulation
- papilla base (Experimental): Strangulation is applied on the the buccal side of the attached gingiva, on the base of the mesial papilla of tooth 12, in straight line going from one side of papilla to the other.
  Interventions: Procedure: strangulation

INTERVENTIONS:
Procedure: strangulation — The strangulation is applied on the attached gingiva with an angulated manual instrument. The force of the occlusion is standardized by a calibrated spring connecting the head with the handle of the tool. The head is overlaid onto the gingiva covering 10mm long and 1mm width surface. The amount of the applied pressure is 100 gram.

SUMMARY:
Apply the LASCA for follow-up the postocclusive microcirculation after strangulation of the gingiva in order to characterize the kinetics of the blood flow changes in human subjects.

DETAILED DESCRIPTION:
During surgical endodontics the cortical bone is exposed by elevating a full- thickness tissue flap. Cutting across mucosal blood vessels disturbs perfusion and causes ischemia. On the other hand, preserving sufficient blood flow of the soft tissue segment is important for the postoperative wound healing. In order to minimize the damage of the microvasculature of the operated area, the incision should be properly designed.

The investigators will model surgical incisions by strangulation of the gingiva of healthy human subjects based on the commonly applied endodontic incision such as horizontal, vertical and papilla base. The primary aim is to determine the effect of a short term disruption of the blood flow at the respective region on the surrounding area in order to assess the functionally active collateral circulation. Using Laser Speckle Contrast Analysis (LASCA), which provides blood perfusion data, the investigators will have the possibility to detect functional alterations in gingival microcirculation during and after a short term of strangulation. The secondary aim is to assess the time course of the restoration of the circulation on the affected area.

ELIGIBILITY:
Inclusion Criteria:

* general good health

Exclusion Criteria:

* pregnancy
* smoking
* general diseases
* medicine taking except contraceptives

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2015-10; Primary Completion 2016-02 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in blood flow during and after ischemia | baseline, at time of strangulation, and 30 second, 5,10,15,20 minute post-occlusal
  The blood flow changes are measured by Laser Speckle Contrast Analyzer (LASCA) before (baseline), during and after strangulation. The scale is an arbitrary unit (0-3000 LSPU) and the relative changes to the baseline measurement will be calculate. The blood flow is recorded for 30min.